CLINICAL TRIAL: NCT01882439
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study Of The Efficacy And Safety Of 2 Doses Of Tofacitinib (Cp-690,550) In Subjects With Active Psoriatic Arthritis And An Inadequate Response To At Least One Tnf Inhibitor
Brief Title: Tofacitinib In Psoriatic Arthritis Subjects With Inadequate Response to TNF Inhibitors
Acronym: OPAL BEYOND
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A3921125; 2013-001368-46 (EudraCT Number)
Record Dates: First submitted 2013-06-18; First posted 2013-06-20 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Psoriatic Arthritis
Keywords: psoriatic arthritis; tofacitinib; ACR20; HAQ-DI; TNF inhibitor failure
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — tofacitinib

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Treatment Sequence A (Experimental): Tofacitinib 5 mg BID for 6 months
  Interventions: Drug: Tofacitinib
- Treatment Sequence B (Experimental): Tofacitinib 10 mg BID for 6 months
  Interventions: Drug: Tofacitinib
- Treatment Sequence C (Placebo Comparator): Placebo for 3 months then tofacitinib 5 mg BID for 3 months
  Interventions: Other: Placebo; Drug: Tofacitinib
- Treatment Sequence D (Placebo Comparator): Placebo for 3 months then tofacitinib 10 mg BID for 3 months
  Interventions: Other: Placebo; Drug: Tofacitinib

INTERVENTIONS:
Drug: Tofacitinib — tablets, 5 mg BID x 6 months
  Arms: Treatment Sequence A
Drug: Tofacitinib — tablets, 10 mg BID x 6 months
  Arms: Treatment Sequence B
Other: Placebo — tablets, to match tofacitinib 5 mg BID x 3 months
  Arms: Treatment Sequence C
Drug: Tofacitinib — tablets, 5 mg BID x 3 months
  Arms: Treatment Sequence C
Other: Placebo — tablets, to match tofacitinib 10 mg BID x 3 months
  Arms: Treatment Sequence D
Drug: Tofacitinib — tablets, 10 mg BID x 3 months
  Arms: Treatment Sequence D

SUMMARY:
To examine the safety and efficacy of tofacitinib in subjects with active psoriatic arthritis who have previously had an inadequate response to at least one TNF inhibitor either due to lack of efficacy or an adverse event.

ELIGIBILITY:
Inclusion Criteria:

* Active arthritis at screening/baseline as indicated by >/= 3 tender/painful and 3 swollen joints
* Active plaque psoriasis at screening
* Inadequate efficacy or lack of toleration to previously administered TNF inhibitor

Exclusion Criteria:

* Non-plaque forms of psoriasis (with exception of nail psoriasis)
* History of autoimmune rheumatic disease other than PsA; also prior history of or current, rheumatic inflammatory disease other than PsA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (125):
- United States (43):
  - Rheumatology Associates P.C., Birmingham, Alabama
  - Rheumatology Associates of North Alabama, PC, Huntsville, Alabama
  - Arizona Arthritis & Rheumatology Associates, P.C., Glendale, Arizona
  - Medvin Clinical Research, Covina, California
  - St. Jude Hospital Yorba Linda DBA St. Joseph Heritage Healthcare, Fullerton, California
  - Ronald Reagan UCLA Medical Center, Drug Information Center, Los Angeles, California
  - UCLA David Geffen School of Medicine, Los Angeles, California
  - San Diego Arthritis Medical Clinic, San Diego, California
  - Stanford Hospital and Clinics, Stanford, California
  - New England Research Associates, LLC, Trumbull, Connecticut
  - Rheumatology Associates of Central Florida, PA, Orlando, Florida
  - Millennium Research, Ormond Beach, Florida
  - Arthritis Center, Inc., Palm Harbor, Florida
  - Integral Rheumatology & Immunology Specialists (IRIS), Plantation, Florida
  - Florida Medical Clinic, P.A., Zephyrhills, Florida
  - St. Luke's Clinic - Rheumatology, Boise, Idaho
  - St. Luke's Intermountain Research Center, Boise, Idaho
  - Bluegrass Community Research, Inc, Lexington, Kentucky
  - Klein & Associates, M.D., P.A., Hagerstown, Maryland
  - The Center For Rheumatology And Bone Research, Wheaton, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Clinical Pharmacology Study Group, Worcester, Massachusetts
  - St. Paul Rheumatology, PA, Eagan, Minnesota
  - Clayton Medical Research, St Louis, Missouri
  - Physician Research Collaboration, LLC, Lincoln, Nebraska
  - Dartmouth-Hitchcock Medical Center (DHMC), Lebanon, New Hampshire
  - Cincinnati Rheumatic Disease Study Group, Inc., Cincinnati, Ohio
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - Paramount Medical Research & Consulting, LLC, Middleburg Heights, Ohio
  - East Penn Rheumatology Associates, PC, Bethlehem, Pennsylvania
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
  - Low Country Rheumatology, PA, Charleston, South Carolina
  - Arthritis Clinic, Jackson, Tennessee
  - West Tennessee Research Institute, Jackson, Tennessee
  - Adriana M. Pop-Moody, M.D., Clinic, P.A., Corpus Christi, Texas
  - Pioneer Research Solutions, Inc., Cypress, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Drug Shipment/Storage: Investigational Drug Services, Salt Lake City, Utah
  - University of Utah Hospital & Clinics, Salt Lake City, Utah
  - Dynacare Laboratories, Seattle, Washington
  - Seattle Rheumatology Associates, Seattle, Washington
  - Swedish Medical Center, Seattle, Washington
- Australia (3):
  - Royal Prince Alfred Hospital, Rheumatology Department, Camperdown, New South Wales
  - Rheumatology Research Unit, Maroochydore, Queensland
  - Emeritus Research Pty Ltd, Malvern East, Victoria
- Belgium (5):
  - Hospital Erasme - Clinique Universitaire de Bruxelles, Brussels
  - ReumaClinic, Genk
  - Universitair Ziekenhuis Gent, Ghent
  - University Hospital Leuven, Department of Rheumatology, Leuven
  - ZNA Jan Palfijn, Merksem
- Brazil (6):
  - CMIP: Centro Mineiro de Pesquisa Ltda /, Juiz de Fora, Minas Gerais
  - CETAC - DIAGNOSTICO POR IMAGEM (image only), Curitiba, Paraná
  - EDUMED - Educacao em Saude SS LTDA., Curitiba, Paraná
  - Hospital de Clinicas de Porto Alegre (HCPA) / UFRGS, Porto Alegre, Rio Grande do Sul
  - Clinica Medica Bonfiglioli Ltda. / Clinica Bonfiglioli, Campinas, São Paulo
  - Radiologia Clínica de Campinas - RCC (Images only), Campinas, São Paulo
- Medical Plus s.r.o., Uherské Hradiště, Czechia
- France (2):
  - Centre Hospitalier Sud-Francilien - Secretariat de Rhumatologie, Corbeil-Essonnes, Cedex
  - Hopital Avicenne, Bobigny
- Germany (10):
  - Rheumazentrum Prof. Dr. med Gunther Neeck, Bad Doberan
  - Charite Universitatsmedizin Berlin - Campus Charite Mitte, Berlin
  - Rheumapraxis Steglitz, Berlin
  - Schlosspark-Klinik, Berlin
  - University Hospital of Cologne, Cologne
  - Universitaetsklinikum Erlangen, Medizinische Klinik 3, Erlangen
  - CIRI - Centrum für innovative Diagnostik und Therapie Rheumatologie/Immunologie (GmbH), Frankfurt am Main
  - Medizinische Universitatsklinik Freiburg, Freiburg im Breisgau
  - Universitaetsklinikum Des Saarlandes Und Medizinische Fakultaet Der Universitaet Des Saarlandes, Homburg
  - Elisabeth Klinik Bigge, Olsberg
- Mexico (18):
  - Hospital Angeles Clinica Londres, Mexico City, D.F
  - Centro Integral en Reumatologia SA de CV, Guadalajara, Jalisco
  - Grupo Santa Bernardette S.A. de C.V., Guadalajara, Jalisco
  - Grupo Medico Camino S.C., Mexico City, Mexico City
  - CLIDITER, S.A. de C.V., Mexico City, Mexico City
  - Universidad La Salle AC, Mexico City, Mexico City
  - Medica Sur, S.A.B. de C.V. (For Emergencies Only), Mexico City, Mexico City
  - Centro de Investigacion de Tratamientos Innovadores de Sinaloa, S.C, Culiacán, Sinaloa
  - Sanatorio CEMSI Chapultepec (For Emergencies Only), Culiacán, Sinaloa
  - Hospital General de Culiacan "Dr. Bernardo J. Gastelum", Culiacán, Sinaloa
  - Star Medica S.A. de C.V. (For Emergencies Only), Merdia, Yucatán
  - Institute Medico Panamericano, S.A. de C.V. (For Emergencies Only), Mérida, Yucatán
  - Unidad Reumatologica Las Americas SCP, Mérida, Yucatán
  - Centro de Investigacion Clinica Pensiones, Mérida, Yucatán
  - Centro Multidisciplinario para el Desarrollo, Mérida, Yucatán
  - Hospital Star Medica Merida (For Emergencies Only), Mérida, Yucatán
  - Christus Muguerza del parque, S.A de C.V, Chihuahua City
  - Investigacion y Biomedicina de Chihuahua, Chihuahua City
- Poland (9):
  - Centrum Kliniczno-Badawcze J.Brzezicki, B.Gornikiewicz-Brzez, Elblag
  - Centrum Radiologii for X-Ray only, Elblag
  - NZOZ Centrum Reumatologiczne Indywidualna Specjalistyczna Praktyka Lekarska Lek. Med. Barbara Bazela, Elblag
  - Wojewodzki Szpital Zespolony Zaklad Radiologii, Elblag
  - Przychodnia Specjalistyczna Lekarskiej Spozielni Pracy "Medica" for X-Ray Only, Grodzisk Mazowiecki
  - Specjalistyczne Gabinety Lekarskie "DERMED" Anna Kaszuba, Lodz
  - NZOZ Lecznica MAK-MED S.C., Nadarzyn
  - Prywatna Praktyka Lekarska Prof. UM dr hab. Pawel Hrycaj, Poznan
  - Reumatika Centrum Reumatologii nzoz, Warsaw
- Russia (7):
  - Regional State Budgetary Healthcare Institution of Karelia Republic "Republic Hospital n.a., Petrozavodsk, Karelia Republic
  - State Autonomic Healthcare Institution City Clinical Hospital # 7, Kazan', Republic of Tatarstan, Russia
  - SBIH of Moscow "City Clinical Hospital#1 n. a. N.I. Pirogov" of the Healthcare Department of Moscow, Moscow
  - City Neurological Centre "SibNeyroMed", LLC, Novosibirsk
  - Limited Liability Company Consultative Diagnostic Rheumatology Center "Healthy Joints", Novosibirsk
  - State Budget Educational Institution of Highest Professional Education, Tomsk
  - State Institution of Healthcare of Yaroslavl Region, Yaroslavl
- MEDMAN s.r.o. - reumatologicka ambulancia, Martin, Slovakia
- Spain (8):
  - Hospital Clinico de Santiago, Santiago de Compostela, A Coruna
  - Corporacio Sanitaria Parc Tauli, Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla, Santander, Cantabria
  - Hospital Sierrallana, Torrelavega, Cantabria
  - Complejo Hospitalario Universitario A Coruna, A Coruña
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitaro Y Politecnico La Fe, Valencia
- Taiwan (5):
  - Taipei Veterans General Hospital, Taipei, Taiwan Roc
  - Buddhist Dalin Tzu Chi General Hospital, Chiayi City
  - Chang Gung Medical Foundation-Kaohsiung Branch, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - China Medical University Hospital, Taichung
- United Kingdom (7):
  - Barking Havering and Redbridge University Hospitals NHS Trust, Goodmayes, Essex
  - Barking, Havering and Redbridge University Hospitals NHS Trust, Romford, Essex
  - The Dudley Group NHS Foundation Trust, Dudley, West Midlands
  - Bradford Royal Infirmary, BTHFT, Bradford, West Yorkeshire
  - Royal United Hospitals NHS Foundation Trust, Bath
  - Bradford Teaching Hospitals NHS Foundation Trust, Bradford
  - York Hospital, York Teaching Hospital NHS Foundation Trust, York

REFERENCES:
- [Derived] Gossec L, Sellas A, Gruben DC, Valderrama M, Gomez S, Kinch C, Citera G. Response to Tofacitinib in Patients with Psoriatic Arthritis and Probable Anxiety/Depressive Disorder: A Post Hoc Analysis of Phase 3 Trials. Rheumatol Ther. 2025 Dec;12(6):1175-1186. doi: 10.1007/s40744-025-00800-7. Epub 2025 Oct 28. PMID 41148555
- [Derived] Gladman D, Tillett W, Gruben D, Coates LC, Hahne S, Volkov M. Identification of distinct disease activity trajectories in patients with psoriatic arthritis receiving tofacitinib: a post hoc analysis of two phase 3 studies. RMD Open. 2025 Jun 3;11(2):e005250. doi: 10.1136/rmdopen-2024-005250. PMID 40461265
- [Derived] Gladman DD, Dougados M, Marzo-Ortega H, Cadatal MJ, Agarwal E, Kinch CD, Nash P. Long-term tofacitinib efficacy and safety in psoriatic arthritis with or without prior biologic DMARD exposure: a post hoc analysis. Rheumatol Adv Pract. 2025 Jan 21;9(2):rkaf008. doi: 10.1093/rap/rkaf008. eCollection 2025. PMID 40241921
- [Derived] Mease PJ, Orbai AM, FitzGerald O, Bedaiwi M, Dona L Fleishaker, Mundayat R, Young P, Helliwell PS. Efficacy of tofacitinib on enthesitis in patients with active psoriatic arthritis: analysis of pooled data from two phase 3 studies. Arthritis Res Ther. 2023 Aug 22;25(1):153. doi: 10.1186/s13075-023-03108-5. PMID 37608391
- [Derived] Eder L, Gladman DD, Mease P, Pollock RA, Luna R, Aydin SZ, Ogdie A, Polachek A, Gruben D, Cadatal MJ, Kinch C, Strand V. Sex differences in the efficacy, safety and persistence of patients with psoriatic arthritis treated with tofacitinib: a post-hoc analysis of phase 3 trials and long-term extension. RMD Open. 2023 Mar;9(1):e002718. doi: 10.1136/rmdopen-2022-002718. PMID 36958766
- [Derived] Kristensen LE, Danese S, Yndestad A, Wang C, Nagy E, Modesto I, Rivas J, Benda B. Identification of two tofacitinib subpopulations with different relative risk versus TNF inhibitors: an analysis of the open label, randomised controlled study ORAL Surveillance. Ann Rheum Dis. 2023 Jul;82(7):901-910. doi: 10.1136/ard-2022-223715. Epub 2023 Mar 17. PMID 36931693
- [Derived] Dougados M, Taylor PC, Bingham CO 3rd, Fallon L, Brault Y, Roychoudhury S, Wang L, Kessouri M. The effect of tofacitinib on residual pain in patients with rheumatoid arthritis and psoriatic arthritis. RMD Open. 2022 Sep;8(2):e002478. doi: 10.1136/rmdopen-2022-002478. PMID 36814062
- [Derived] Winthrop KL, Yndestad A, Henrohn D, Danese S, Marsal S, Galindo M, Woolcott JC, Jo H, Kwok K, Shapiro AB, Jones TV, Diehl A, Su C, Panes J, Cohen SB. Influenza Adverse Events in Patients with Rheumatoid Arthritis, Ulcerative Colitis, or Psoriatic Arthritis in the Tofacitinib Clinical Development Programs. Rheumatol Ther. 2023 Apr;10(2):357-373. doi: 10.1007/s40744-022-00507-z. Epub 2022 Dec 17. PMID 36526796
- [Derived] Schneeberger EE, Citera G, Nash P, Smolen JS, Mease PJ, Soriano ER, Helling C, Szumski AE, Mundayat R, de Leon DP. Comparison of disease activity index for psoriatic arthritis (DAPSA) and minimal disease activity (MDA) targets for patients with psoriatic arthritis: A post hoc analysis of data from phase 3 tofacitinib studies. Semin Arthritis Rheum. 2023 Feb;58:152134. doi: 10.1016/j.semarthrit.2022.152134. Epub 2022 Nov 13. PMID 36476498
- [Derived] de Vlam K, Mease PJ, Bushmakin AG, Fleischmann R, Ogdie A, Azevedo VF, Merola JF, Woolcott J, Cappelleri JC, Fallon L, Taylor PC. Identifying and Quantifying the Role of Inflammation in Pain Reduction for Patients With Psoriatic Arthritis Treated With Tofacitinib: A Mediation Analysis. Rheumatol Ther. 2022 Oct;9(5):1451-1464. doi: 10.1007/s40744-022-00482-5. Epub 2022 Sep 8. PMID 36076054
- [Derived] Orbai AM, Mease PJ, Helliwell PS, FitzGerald O, Fleishaker DL, Mundayat R, Young P. Effect of tofacitinib on dactylitis and patient-reported outcomes in patients with active psoriatic arthritis: post-hoc analysis of phase III studies. BMC Rheumatol. 2022 Sep 1;6(1):68. doi: 10.1186/s41927-022-00298-4. PMID 36045453
- [Derived] Taylor PC, Bushmakin AG, Cappelleri JC, Young P, Germino R, Merola JF, Yosipovitch G. Relationships of dermatologic symptoms and quality of life in patients with psoriatic arthritis: analysis of two tofacitinib phase III studies. J Dermatolog Treat. 2022 Aug;33(5):2614-2620. doi: 10.1080/09546634.2022.2060924. Epub 2022 Apr 11. PMID 35385361
- [Derived] Gladman DD, Coates LC, Wu J, Fallon L, Bacci ED, Cappelleri JC, Bushmakin AG, Helliwell PS. Time to response for clinical and patient-reported outcomes in patients with psoriatic arthritis treated with tofacitinib, adalimumab, or placebo. Arthritis Res Ther. 2022 Feb 9;24(1):40. doi: 10.1186/s13075-022-02721-0. PMID 35139908
- [Derived] Dikranian A, Gold D, Bessette L, Nash P, Azevedo VF, Wang L, Woolcott J, Shapiro AB, Szumski A, Fleishaker D, Wollenhaupt J. Frequency and Duration of Early Non-serious Adverse Events in Patients with Rheumatoid Arthritis and Psoriatic Arthritis Treated with Tofacitinib. Rheumatol Ther. 2022 Apr;9(2):411-433. doi: 10.1007/s40744-021-00405-w. Epub 2021 Dec 17. PMID 34921355
- [Derived] Winthrop KL, Curtis JR, Yamaoka K, Lee EB, Hirose T, Rivas JL, Kwok K, Burmester GR. Clinical Management of Herpes Zoster in Patients With Rheumatoid Arthritis or Psoriatic Arthritis Receiving Tofacitinib Treatment. Rheumatol Ther. 2022 Feb;9(1):243-263. doi: 10.1007/s40744-021-00390-0. Epub 2021 Dec 6. PMID 34870800
- [Derived] Kivitz AJ, FitzGerald O, Nash P, Pang S, Azevedo VF, Wang C, Takiya L. Efficacy and safety of tofacitinib by background methotrexate dose in psoriatic arthritis: post hoc exploratory analysis from two phase III trials. Clin Rheumatol. 2022 Feb;41(2):499-511. doi: 10.1007/s10067-021-05894-2. Epub 2021 Sep 12. PMID 34510295
- [Derived] de Vlam K, Ogdie A, Bushmakin AG, Cappelleri JC, Fleischmann R, Taylor PC, Azevedo V, Fallon L, Woolcott J, Mease PJ. Median time to pain improvement and the impact of baseline pain severity on pain response in patients with psoriatic arthritis treated with tofacitinib. RMD Open. 2021 Jul;7(2):e001609. doi: 10.1136/rmdopen-2021-001609. PMID 34226183
- [Derived] Coates LC, Bushmakin AG, FitzGerald O, Gladman DD, Fallon L, Cappelleri JC, Hsu MA, Helliwell PS. Relationships between psoriatic arthritis composite measures of disease activity with patient-reported outcomes in phase 3 studies of tofacitinib. Arthritis Res Ther. 2021 Mar 26;23(1):94. doi: 10.1186/s13075-021-02474-2. PMID 33766074
- [Derived] Ritchlin CT, Giles JT, Ogdie A, Gomez-Reino JJ, Helliwell P, Young P, Wang C, Wu J, Romero AB, Woolcott J, Stockert L. Tofacitinib in Patients With Psoriatic Arthritis and Metabolic Syndrome: A Post hoc Analysis of Phase 3 Studies. ACR Open Rheumatol. 2020 Oct;2(10):543-554. doi: 10.1002/acr2.11166. Epub 2020 Sep 10. PMID 32910531
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Burmester GR, Curtis JR, Yun H, FitzGerald O, Winthrop KL, Azevedo VF, Rigby WFC, Kanik KS, Wang C, Biswas P, Jones T, Palmetto N, Hendrikx T, Menon S, Rojo R. An Integrated Analysis of the Safety of Tofacitinib in Psoriatic Arthritis across Phase III and Long-Term Extension Studies with Comparison to Real-World Observational Data. Drug Saf. 2020 Apr;43(4):379-392. doi: 10.1007/s40264-020-00904-9. PMID 32006348
- [Derived] Gladman DD, Charles-Schoeman C, McInnes IB, Veale DJ, Thiers B, Nurmohamed M, Graham D, Wang C, Jones T, Wolk R, DeMasi R. Changes in Lipid Levels and Incidence of Cardiovascular Events Following Tofacitinib Treatment in Patients With Psoriatic Arthritis: A Pooled Analysis Across Phase III and Long-Term Extension Studies. Arthritis Care Res (Hoboken). 2019 Oct;71(10):1387-1395. doi: 10.1002/acr.23930. PMID 31112005
- [Derived] Cella D, Wilson H, Shalhoub H, Revicki DA, Cappelleri JC, Bushmakin AG, Kudlacz E, Hsu MA. Content validity and psychometric evaluation of Functional Assessment of Chronic Illness Therapy-Fatigue in patients with psoriatic arthritis. J Patient Rep Outcomes. 2019 May 20;3(1):30. doi: 10.1186/s41687-019-0115-4. PMID 31111255
- [Derived] Strand V, de Vlam K, Covarrubias-Cobos JA, Mease PJ, Gladman DD, Chen L, Kudlacz E, Wu J, Cappelleri JC, Hendrikx T, Hsu MA. Effect of tofacitinib on patient-reported outcomes in patients with active psoriatic arthritis and an inadequate response to tumour necrosis factor inhibitors in the phase III, randomised controlled trial: OPAL Beyond. RMD Open. 2019 Jan 11;5(1):e000808. doi: 10.1136/rmdopen-2018-000808. eCollection 2019. PMID 30713722
- [Derived] Cella D, Wilson H, Shalhoub H, Revicki DA, Cappelleri JC, Bushmakin AG, Kudlacz E, Hsu MA. Content validity and psychometric evaluation of Functional Assessment of Chronic Illness Therapy-Fatigue in patients with psoriatic arthritis. J Patient Rep Outcomes. 2019 Jan 24;3(1):5. doi: 10.1186/s41687-019-0094-5. PMID 30680661 (Retraction: PMID 31139969 J Patient Rep Outcomes. 2019 May 28;3(1):32)
- [Derived] Nash P, Coates LC, Fleischmann R, Papp KA, Gomez-Reino JJ, Kanik KS, Wang C, Wu J, Menon S, Hendrikx T, Ports WC. Efficacy of Tofacitinib for the Treatment of Psoriatic Arthritis: Pooled Analysis of Two Phase 3 Studies. Rheumatol Ther. 2018 Dec;5(2):567-582. doi: 10.1007/s40744-018-0131-5. Epub 2018 Nov 9. PMID 30414064
- [Derived] Helliwell P, Coates LC, FitzGerald O, Nash P, Soriano ER, Elaine Husni M, Hsu MA, Kanik KS, Hendrikx T, Wu J, Kudlacz E. Disease-specific composite measures for psoriatic arthritis are highly responsive to a Janus kinase inhibitor treatment that targets multiple domains of disease. Arthritis Res Ther. 2018 Oct 29;20(1):242. doi: 10.1186/s13075-018-1739-0. PMID 30373651
- [Derived] Gladman D, Rigby W, Azevedo VF, Behrens F, Blanco R, Kaszuba A, Kudlacz E, Wang C, Menon S, Hendrikx T, Kanik KS. Tofacitinib for Psoriatic Arthritis in Patients with an Inadequate Response to TNF Inhibitors. N Engl J Med. 2017 Oct 19;377(16):1525-1536. doi: 10.1056/NEJMoa1615977. PMID 29045207
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921125&StudyName=Tofacitinib%20In%20Psoriatic%20Arthritis%20Subjects%20With%20Inadequate%20Response%20to%20TNF%20Inhibitors

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data through End of Study (Month 6)
Pre-assignment Details: Of 546 participants screened for entry into the study, 395 were enrolled and randomized, 394 received treatment.
Groups:
- Tofacitinib, 5 mg Twice Daily: Participants received one 5 mg tofacitinib tablet, twice daily, and one placebo tablet twice daily.
- Tofacitinib, 10 mg, Twice Daily: Participants received two 5 mg tofacitinib tablets, twice daily.
- Placebo/Tofacitinib, 5 mg, Twice Daily: Participants received two placebo tablets, twice daily, up to 3 months. At the end of this period, participants received one 5 mg tofacitinib tablet, twice daily, and one placebo tablet, twice daily.
- Placebo/Tofacitinib, 10 mg, Twice Daily: Participants received two placebo tablets, twice daily, up to 3 months. At the end of this period, participants received two 5 mg tofacitinib tablets, twice daily.
Period: Overall Study
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily
Started | 131 (Received treatment) | 132 (Received treatment) | 66 (Received treatment) | 65 (Received treatment)
Completed | 122 | 111 | 56 | 56
Not Completed | 9 | 21 | 10 | 9
Not completed — Adverse event related to study drug | 3 | 8 | 1 | 2
Not completed — Pregnancy | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 2 | 2 | 0 | 1
Not completed — No longer willing to participate | 1 | 4 | 2 | 3
Not completed — Medication error with no associated AE | 0 | 0 | 2 | 0
Not completed — Insufficient clinical response | 1 | 4 | 4 | 2
Not completed — Adverse event unrelated to study drug | 2 | 2 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Total
Number analyzed (Participants) | 131 | 132 | 66 | 65 | 394
Age, Continuous [Mean (Standard Deviation); unit: Years] | 49.5 (12.3) | 51.3 (10.9) | 48.7 (11.2) | 49.3 (14.0) | 50.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 74 | 38 | 42 | 218
  Male | 67 | 58 | 28 | 23 | 176

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Meeting American College of Rheumatology Response Criteria Greater Than or Equal to (≥) 20% (ACR20): Month 3
Description: ACR20 was calculated as a ≥20% improvement from baseline in tender/painful and swollen joint counts and ≥20% improvement from baseline in 3 of the 5 remaining ACR core set measures: patient's global assessment of arthritis, physician's global assessment of arthritis, patient's assessment of arthritis pain, Health Assessment Questionnaire - Disability Index (HAQ-DI), and C-reactive protein (CRP).
Time Frame: Month 3
Population: All participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Tofacitinib, 5 mg Twice Daily: Participants received one 5 mg tofacitinib tablet twice daily and one placebo tablet twice daily.
- Tofacitinib, 10 mg, Twice Daily: Participants received two 5 mg tofacitinib tablets twice daily.
- Placebo: Participants received two placebo tablets twice daily up to 3 months.
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 131 | 132 | 131
Percentage of participants | 49.62 [14.72 to 37.19] | 46.97 [12.10 to 34.51] | 23.66 [-14.72 to 9.43]
Statistical Analysis 1: Comparison: Tofacitinib, 5 mg Twice Daily vs Placebo; Test type: Superiority or Other; p < 0.0001, Large sample approximation; Missing response (MR) = non-response (NR); Risk Difference (RD) = 25.95, 95% CI 2-sided [14.72 to 37.19], Standard Error of Mean 5.73
Statistical Analysis 2: Comparison: Tofacitinib, 10 mg, Twice Daily vs Placebo; Test type: Superiority or Other; p < 0.0001, Large sample approximation; MR=NR; Risk Difference (RD) = 23.31, 95% CI 2-sided [12.10 to 34.51], Standard Error of Mean 5.71

2. Primary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score: Month 3
Description: The HAQ-DI assesses the difficulty a patient has had in the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2-3 items. For each question, level of difficulty is scored from 0 to 3 with 0=no difficulty, 1=some difficulty, 2=much difficulty, and 3=unable to do. The score for each domain is the maximum (worst) score from the items/questions within the domain. Higher score indicates greater disability. Overall score was computed as the sum of the domain scores divided by the number of domains answered. The total possible score ranged from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability.
Time Frame: Month 3
Population: All participants who were randomized, received at least 1 dose of study drug, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 129 | 132 | 131
Units on a scale | -0.3920 (0.04544) | -0.3540 (0.04579) | -0.1391 (0.04573)
Statistical Analysis 1: Comparison: Tofacitinib, 5 mg Twice Daily vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed Models Analysis; No imputation; Mean Difference (Net) = -0.2529, 95% CI 2-sided [-0.3792 to -0.1266], Standard Error of Mean 0.06422
Statistical Analysis 2: Comparison: Tofacitinib, 10 mg, Twice Daily vs Placebo; Test type: Superiority or Other; p = 0.0009, Mixed Models Analysis; No imputation; Mean Difference (Net) = -0.2150, 95% CI 2-sided [-0.3419 to -0.0881], Standard Error of Mean 0.06453

3. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology Response Criteria ≥50% (ACR50) at Week 2 and Months 1, 2, 3, 4, and 6
Description: ACR50 was calculated as a ≥50% improvement from baseline in tender /painful and swollen joint counts and ≥50% improvement from baseline in 3 of the 5 remaining ACR core set measures: patient's global assessment of arthritis, physician's global assessment of arthritis, patient's assessment of arthritis pain, HAQ-DI, and CRP. n=number of responders.
Time Frame: Week 2 and Months 1, 2, 3, 4, and 6
Population: All participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo/Tofacitinib, 5 mg, Twice Daily: Participants received two placebo tablets twice daily up to 3 months. At the end of this period, participants received one 5 mg tofacitinib tablet twice daily and one placebo tablet twice daily.
- Placebo/Tofacitinib, 10 mg, Twice Daily: Participants received two placebo tablets twice daily up to 3 months. At the end of this period, participants received two 5 mg tofacitinib tablet twice daily.
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 131 | 132 | 66 | 65 | 131
Percentage of participants
  Week 2 (n=8,13,NA,NA,4) | 6.11 | 9.85 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 3.05
  Month 1 (n=23,14,NA,NA,8) | 17.56 | 10.61 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 6.11
  Month 2 (n=33,30,NA,NA,14) | 25.19 | 22.73 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 10.69
  Month 3 (n=39,37,NA,NA,19) | 29.77 | 28.03 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 14.50
  Month 4 (n=50,38,15,21,NA) | 38.17 | 28.79 | 22.73 | 32.31 | NA — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.
  Month 6 (n=50,39,21,23,NA) | 38.17 | 29.55 | 31.82 | 35.38 | NA — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

4. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology Response Criteria ≥70% (ACR70) at Week 2 and Months 1, 2, 3, 4, and 6
Description: ACR70 was calculated as a ≥70% improvement from baseline in tender /painful and swollen joint counts and ≥70% improvement from baseline in 3 of the 5 remaining ACR core set measures: patient's global assessment of arthritis, physician's global assessment of arthritis, patient's assessment of arthritis pain, HAQ-DI, and CRP. n=number of responders.
Time Frame: Week 2 and Months 1, 2, 3, 4, and 6
Population: All participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Groups:
- Placebo/Tofacitinib, 5 mg, Twice Daily: Participants received two placebo tablets twice daily for 3 months. At the end of this period, participants received one 5 mg tofacitinib tablet twice daily and one placebo tablet twice daily.
- Placebo/Tofacitinib, 10 mg, Twice Daily: Participants received two placebo tablets twice daily up to 3 months. At the end of this period, participants received two 5 mg tofacitinib tablets twice daily.
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 131 | 132 | 66 | 65 | 131
Percentage of participants
  Week 2 (n=2,3,NA,NA,1) | 1.53 | 2.27 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 0.76
  Month 1 (n=7,5,NA,NA,3) | 5.34 | 3.79 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.29
  Month 2 (n=17,13,NA,NA,6) | 12.98 | 9.85 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 4.58
  Month 3 (n=22,19,NA,NA,13) | 16.79 | 14.39 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 9.92
  Month 4 (n=24,20,6,14,NA) | 18.32 | 15.15 | 9.09 | 21.54 | NA — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.
  Month 6 (n=28,19,10,12,NA) | 21.37 | 14.39 | 15.15 | 18.46 | NA — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

5. Secondary Outcome: Percentage of Participants Meeting American College of Rheumatology Response Criteria Greater Than or Equal to (≥) 20% (ACR20): Week 2 and Months 1, 2, 4, and 6
Description: ACR20 was calculated as a ≥20% improvement from baseline in tender /painful and swollen joint counts and ≥20% improvement from baseline in 3 of the 5 remaining ACR core set measures: patient's global assessment of arthritis, physician's global assessment of arthritis, patient's assessment of arthritis pain, HAQ-DI, and CRP. n=number of responders.
Time Frame: Week 2 and Months 1, 2, 4, and 6
Population: All participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 131 | 132 | 66 | 65 | 131
Percentage of participants
  Week 2 (n=35,38,NA,NA,17) | 26.72 | 28.79 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 12.98
  Month 1 (n=45,56,NA,NA,29) | 34.35 | 42.42 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 22.14
  Month 2 (n=63,63,NA,NA,34) | 48.09 | 47.73 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 25.95
  Month 4 (n=78,69,30,33,NA) | 59.54 | 52.27 | 45.45 | 50.77 | NA — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.
  Month 6 (n=78,65,33,35,NA) | 59.54 | 49.24 | 50.00 | 53.85 | NA — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

6. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) Score: Week 2 and Months 1, 2, 4, and 6
Description: The HAQ-DI assesses the difficulty a patient has had in the past week in 8 domains of daily living activities: dressing and grooming, arising, eating, walking, hygiene, reach, grip, and other activities. Each activity category consists of 2-3 items. For each question, level of difficulty is scored from 0 to 3 with 0=no difficulty, 1=some difficulty, 2=much difficulty, and 3=unable to do. The score for each domain is the maximum (worst) score from the items/questions within the domain. Higher score indicates greater disability. Overall score was computed as the sum of the domain scores divided by the number of domains answered. The total possible score ranged from 0 to 3 where 0 = least difficulty and 3 = extreme difficulty. Higher overall score indicates greater disability. n=number of participants evaluable at each visit.
Time Frame: Week 2 and Months 1, 2, 4, and 6
Population: All participants who were randomized, received at least 1 dose of study drug, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 129 | 132 | 66 | 65 | 131
Units on scale
  Week 2 (129,130,NA,NA,128) | -0.2198 (0.03145) | -0.1652 (0.03160) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.0655 (0.03133)
  Month 1 (128,129,NA,NA,130) | -0.3229 (0.04074) | -0.2279 (0.04073) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.1481 (0.04038)
  Month 2 (125,126,NA,NA,121) | -0.4114 (0.04311) | -0.3131 (0.04316) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.1620 (0.04317)
  Month 4 (125,121,57,58,NA) | -0.4455 (0.04489) | -0.3305 (0.04523) | -0.3836 (0.06443) | -0.3918 (0.06418) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.
  Month 6 (122,112,56,56,NA) | -0.4365 (0.04642) | -0.3397 (0.04720) | -0.4808 (0.06680) | -0.4157 (0.06665) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

7. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Response Criteria Components: C-reactive Protein (CRP) Levels: Month 3
Description: The test for CRP is a laboratory measurement for evaluation of an acute phase reactant of inflammation through the use of an ultrasensitive assay. A decrease in the level of CRP indicates reduction in inflammation and therefore improvement.
Time Frame: Month 3
Population: All participants who were randomized, received at least 1 dose of study drug, and were evaluable
Measure: Least Squares Mean (Standard Error); unit: mg/L
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 130 | 132 | 131
mg/L | -5.4657 (1.80096) | -5.9156 (1.83181) | 1.0233 (1.82879)

8. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Response Criteria Components Score: Patient's Assessment of Arthritis Pain: Month 3
Description: Participants assessed the severity of their arthritis pain using a 100 mm visual analog scale (VAS) by placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponded to the magnitude of their pain.
Time Frame: Month 3
Population: All participants who were randomized, received at least 1 dose of study drug, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 129 | 132 | 131
mm | -21.66 (2.162) | -20.88 (2.188) | -7.72 (2.184)

9. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Response Criteria Components Score: Patient's Global Assessment of Arthritis: Month 3
Description: Participants answered the following question, "Considering all the ways your arthritis affects you, how are you feeling today?" The participant's response was recorded using a 100 mm VAS by placing a mark on the scale between 0 (very well) and 100 (very poorly).
Time Frame: Month 3
Population: All participants who were randomized, received at least 1 dose of study drug, and were evaluable
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 129 | 132 | 131
mm | -21.59 (2.228) | -19.88 (2.248) | -7.14 (2.247)

10. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Response Criteria Components Score: Physician's Global Assessment of Arthritis: Month 3
Description: The blinded investigator or qualified assessor assessed how the participant's overall arthritis appeared at the time of the visit. This was an evaluation based on the participant's disease signs, functional capacity and physical examination, and was independent of the Patient's Global Assessment of Arthritis. The investigator's response was recorded using a 100 mm VAS by placing a mark on the scale between 0 (very good) and 100 (very poor).
Time Frame: Month 3
Population: All participants who were randomized, received at least 1 dose of study drug, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 128
mm | -27.25 (1.893) | -28.95 (1.916) | -15.88 (1.929)

11. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Response Criteria Components Score: Swollen Joint Count: Month 3
Description: Swollen joint counts are considered the most specific quantitative clinical measure used to assess the status of participants with inflammatory types of arthritis. Sixty six (66) joints were assessed by a blinded assessor to determine the number of joints that were considered swelling.
Time Frame: Month 3
Population: All participants who were randomized, received at least 1 dose of study drug, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 130 | 132 | 131
Joints | -7.6 (0.59) | -6.7 (0.60) | -2.7 (0.60)

12. Secondary Outcome: Change From Baseline in American College of Rheumatology (ACR) Response Criteria Components Score: Tender/Painful Joint Count: Month 3
Description: Tender/painful joint counts are considered the most specific quantitative clinical measure used to assess the status of participants with inflammatory types of arthritis. Sixty eight (68) joints were assessed by a blinded assessor to determine the number of joints that were considered tender or painful.
Time Frame: Month 3
Population: All participants who were randomized, received at least 1 dose of study drug, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Joints
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 130 | 132 | 131
Joints | -9.9 (0.97) | -9.7 (0.98) | -4.5 (0.98)

13. Secondary Outcome: Percentage of Participants Meeting Psoriatic Arthritis Response Criteria (PsARC): Week 2, Months 1, 2, 3, 4, and 6
Description: The PsARC covers 4 measures: Tender joint count, swollen joint count, the Physician's Global Assessment of Arthritis, and the Patient's Global Assessment of Arthritis. The PsARC response is defined as improvement in 2 of 4 items, 1 of which must be joint pain or swelling, without worsening in any measure. Improvement criteria: ≥20% improvement in Physician's Global Assessment of Arthritis; ≥20% improvement in Patient's Global Assessment of Arthritis; ≥30% improvement in tender joint count; and ≥30% improvement in swollen joint count. n=number of responders.
Time Frame: Week 2, Months 1, 2, 3, 4, and 6
Population: All participants who were randomized and received at least 1 dose of study drug.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 131 | 132 | 66 | 65 | 131
Percentage of participants
  Week 2 (n=43,45,NA,NA,23) | 32.82 | 34.09 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 17.56
  Month 1 (n=56,66,NA,NA,45) | 42.75 | 50.00 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 34.35
  Month 2 (n=67,72,NA,NA,43) | 51.15 | 54.55 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 32.82
  Month 3 (n=77,64,NA,NA,38) | 58.78 | 48.48 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 29.01
  Month 4 (n=74,75,34,38.NA) | 56.49 | 56.82 | 51.52 | 58.46 | NA — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.
  Month 6 (n=77,68,34,36,NA) | 58.78 | 51.52 | 51.52 | 55.38 | NA — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

14. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Psoriasis (PGA-PsO) Response: Months 1, 3, and 6
Description: The PGA-PsO is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are rated separately over the whole body according to a 5-point severity scale, scored as 0=none; 1, 2, 3, or 4=most severe. The severity rating scores are summed and the average taken; the total average is rounded to the nearest whole number score to determine the PGA-PsO score on a scale of 0 to 4 (0=clear, 1=almost clear, 2=mild, 3=moderate, 4=severe). n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, and 6
Population: All participants who were randomized, received at least 1 dose of study drug with baseline PGA-PsO >0, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Groups:
- Tofacitinib, 5 mg Twice Daily; Tofacitinib, 10 mg, Twice Daily: Participants received two 5 mg tofacitinib tablets twice daily.
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 121 | 124 | 63 | 62 | 125
Units on a scale
  Month 1 (n=120,122,NA,NA,125) | -0.5 (0.07) | -0.8 (0.07) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.2 (0.07)
  Month 3 (n=112,116,NA,NA,112) | -0.7 (0.08) | -1.1 (0.08) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.4 (0.08)
  Month 6 (n=116,108,55,51,NA) | -0.9 (0.08) | -1.1 (0.09) | -1.0 (0.12) | -1.0 (0.13) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

15. Secondary Outcome: Percentage of Participants With Psoriasis Area and Severity Index 75 (PASI75) Response: Months 1, 3, and 6
Description: PASI determines psoriasis severity based on lesion severity and percentage of body surface area (BSA) affected. Lesion severity is assessed for erythema, induration, and scaling evaluated separately for the head and neck, upper limbs, trunk, and lower limbs and then rated for each body area according to a 5 point scale: 0=no involvement; 1=slight; 2=moderate; 3=marked; 4=very marked. BSA involvement is the extent (%) of body area affected by psoriasis and is assigned a numerical score: 0=no involvement; 1=0% to 9%; 2=10% to 29%; 3=30% to 49%; 4=50% to 69%; 5=70% to 89%; 6=90% to 100%. In each area, the sum of the severity rating scores is multiplied by the score representing the percentage of this area involved by psoriasis, multiplied by a weighting factor (head 0.1; upper limbs 0.2; trunk 0.3; lower limbs 0.4). The sum of the numbers obtained for each of the 4 body areas is the PASI. PASI75 is defined as a 75% reduction from baseline in PASI. n=number of responders.
Time Frame: Months 1, 3, and 6
Population: All participants who were randomized and received at least 1 dose of study drug with PASI >0 and BSA ≥3% at baseline.
Measure: Number; unit: Percentage of participants
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 80 | 81 | 42 | 44 | 86
Percentage of participants
  Month 1 (n=12,15,NA,NA,5) | 15.00 | 18.52 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 5.81
  Month 3 (n=17,35,NA,NA,12) | 21.25 | 43.21 | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 13.95
  Month 6 (n=27,37,11,14,NA) | 33.75 | 45.68 | 26.19 | 31.82 | NA — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

16. Secondary Outcome: Change From Baseline in Dactylitis Severity Score (DSS): Months 1, 3, and 6
Description: Dactylitis is characterized by swelling of the entire finger or toe. The DSS is a function of finger circumference and tenderness, assessed and summed across all dactylitic digits. The severity of dactylitis is scored on a scale of 0-3, where 0=tenderness and 3=extreme tenderness in each digit of the hands and feet. The range of total dactylitis scores for a participant is 0-60. Higher score indicates greater degree of tenderness. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, and 6
Population: All participants who were randomized, received at least 1 dose of study drug with baseline DSS >0, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 65 | 64 | 29 | 33 | 62
Units on a scale
  Month 1 (n=65,64,NA,NA,62) | -2.8 (0.63) | -4.0 (0.65) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -1.1 (0.64)
  Month 3 (n=64,58,NA,NA,55) | -5.2 (0.73) | -5.4 (0.78) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -1.9 (0.78)
  Month 6 (n=61,55,25,26,NA) | -6.0 (0.84) | -6.0 (0.90) | -5.4 (1.33) | -5.2 (1.26) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

17. Secondary Outcome: Change From Baseline in the Spondyloarthritis Research Consortium of Canada (SPARCC) Enthesitis Index: Months 1, 3, and 6
Description: The SPARCC Enthesitis Index identifies the presence or absence of tenderness at 16 enthesial sites, including the bilateral Achilles tendons, plantar fascia insertion at the calcaneus, patellar tendon insertion at the base of the patella, quadriceps insertion into the superior border of the patella, supraspinatus insertion into the greater tuberosity of the humerus, and medial and lateral epicondyles. On examination, tenderness is recorded as present (1) or absent (0) for each of the 16 sites, with an overall total score ranging from 0 to 16. Higher score indicates a greater number of sites that are affected by enthesitis. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, and 6
Population: All participants who were randomized, received at least 1 dose of study drug with baseline SPARCC Enthesitis Score >0, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units of scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 95 | 105 | 47 | 51 | 98
Units of scale
  Month 1 (n=94,104,NA,NA,98) | -1.9 (0.31) | -1.9 (0.30) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -1.0 (0.30)
  Month 3 (n=92,96,NA,NA,87) | -2.5 (0.34) | -2.8 (0.33) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -1.3 (0.34)
  Month 6 (n=91,93,40,43,NA) | -2.6 (0.36) | -3.1 (0.35) | -2.6 (0.53) | -2.4 (0.51) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

18. Secondary Outcome: Change From Baseline in the Leeds Enthesitis Index (LEI): Months 1, 3, and 6
Description: Enthesitis is inflammation in the tendon, ligament, and joint capsule fiber insertion into bone. The LEI assesses enthesitis in 6 sites. Tenderness is recorded as either present (1) or absent (0) for each of the 6 sites, for a total score of 0-6. Higher score indicates greater severity of enthesitis. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, and 6
Population: All participants who were randomized, received at least 1 dose of study drug with baseline LEI >0, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units of scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 82 | 96 | 45 | 46 | 91
Units of scale
  Month 1 (n=82,95,NA,NA,91) | -1.0 (0.19) | -0.8 (0.18) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.5 (0.18)
  Month 3 (n=79,86,NA,NA,82) | -1.3 (0.19) | -1.3 (0.18) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.5 (0.19)
  Month 6 (n=77,84,38,41,NA) | -1.5 (0.19) | -1.6 (0.18) | -1.4 (0.26) | -1.3 (0.26) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

19. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2, Acute Components (SF-36v2 Acute): Physical Component Summary Score: Months 1, 3, 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The health domains are aggregated into two summary scores known as the physical component summary (PCS) score and the mental component summary (MCS) score. Normalized domain scores, PCS and MCS scores are used in the analyses. The component and domain scores were scored using the United States (US) 1998 general population norms. The resulting norm-based T-scores for both the SF36 version 2 and SF36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher PCS score represents better physical health status. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 124 | 130 | 64 | 65 | 129
T-scores
  Month 1 (n=124,127,NA,NA,129) | 4.65 (0.543) | 3.98 (0.542) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 1.70 (0.534)
  Month 3 (n=121,120,NA,NA,117) | 5.18 (0.684) | 5.34 (0.687) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 1.77 (0.689)
  Month 6 (n=118,110,56,56,NA) | 5.71 (0.751) | 5.00 (0.768) | 6.45 (1.076) | 6.98 (1.074) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

20. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2, Acute Components (SF-36v2 Acute): Mental Component Summary Score: Months 1, 3, 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The health domains are aggregated into two summary scores known as the PCS score and the MCS score. Normalized domain scores, PCS and MCS scores are used in the analyses. The component and domain scores were scored using the US 1998 general population norms. The resulting norm-based T-scores for both the SF36 version 2 and SF36 health domain scales and component summary measures have means of 50 and standard deviations of 10. A higher MCS score represents better mental health status. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 124 | 130 | 64 | 65 | 129
T-scores
  Month 1 (n=124,127,NA,NA,129) | 4.09 (0.740) | 4.19 (0.738) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.33 (0.725)
  Month 3 (n=121,120,NA,NA,117) | 4.94 (0.875) | 4.28 (0.879) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.97 (0.880)
  Month 6 (n=118,110,56,56,NA) | 5.36 (0.878) | 5.37 (0.902) | 5.37 (1.265) | 6.47 (1.259) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

21. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2, Acute Components (SF-36v2 Acute): Physical Functioning Domain: Months 1, 3, 6
Description: SF-36v2 acute is a 36-item measure evaluating 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. The 10 items of the physical functioning scale represent levels & kinds of limitations between extremes of physical activities, including lifting & carrying groceries; climbing stairs; bending, kneeling, or stooping; walking moderate distances; self-care limitations. The physical functioning items capture the presence & extent of physical limitations using a 3-level response continuum. The domain scores were scored using the US 1998 general population norms. The resulting norm-based T-scores for both the SF36 version 2 & SF36 health domain scales & component summary measures have means of 50 & standard deviations of 10. A higher physical functioning domain score represents better physical functioning. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
T-scores
  Month 1 (n=128,129,NA,NA,129) | 3.97 (0.583) | 3.10 (0.587) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 1.55 (0.580)
  Month 3 (n=124,120,NA,NA,117) | 5.00 (0.721) | 4.08 (0.732) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 1.69 (0.734)
  Month 6 (n=121,112,56,56,NA) | 5.39 (0.795) | 3.88 (0.818) | 5.89 (1.153) | 5.60 (1.149) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

22. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2, Acute Components (SF-36v2 Acute): Role-physical Domain: Months 1, 3, 6
Description: SF-36v2 acute is a 36-item measure evaluating 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, & mental health. The 4-item role-physical scale covers an array of physical health-related role limitations, including: a) limitations in the kind of work or other usual activities; b) reductions in the amount of time spent on work or other usual activities; c) difficulty performing work or other usual activities; & d) accomplishing less. Items in the role-physical scale are answered on a 5-point scale. The domain scores were scored using the US 1998 general population norms. The resulting norm-based T-scores for both the SF36 version 2 & SF36 health domain scales & component summary measures have means of 50 & standard deviations of 10. A higher role-physical domain score represents better role-physical functioning. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 126 | 130 | 64 | 65 | 129
T-scores
  Month 1 (n=126,128,NA,NA,129) | 4.22 (0.630) | 3.55 (0.633) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.24 (0.623)
  Month 3 (n=122,120,NA,NA,117) | 4.99 (0.805) | 5.44 (0.814) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.85 (0.814)
  Month 6 (n=120,112,56,56,NA) | 5.58 (0.857) | 5.24 (0.881) | 7.01 (1.241) | 7.21 (1.239) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

23. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2, Acute Components (SF-36v2 Acute): Bodily Pain Domain: Months 1, 3, 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The bodily pain scale comprises of 2 items pertaining to the intensity of bodily pain and extent of interference with normal work activities. The domain scores were scored using the US 1998 general population norms. The resulting norm-based T-scores for both the SF36 version 2 & SF36 health domain scales & component summary measures have means of 50 & standard deviations of 10. A higher bodily pain domain score represents less bodily pain. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 127 | 130 | 64 | 65 | 129
T-scores
  Month 1 (n=127,128,NA,NA,129) | 6.86 (0.634) | 6.39 (0.638) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.31 (0.633)
  Month 3 (n=124,120,NA,NA,117) | 7.00 (0.786) | 7.59 (0.799) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.10 (0.804)
  Month 6 (n=121,112,56,56,NA) | 7.60 (0.848) | 7.69 (0.876) | 8.15 (1.234) | 10.48 (1.236) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

24. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2, Acute Components (SF-36v2 Acute): General Health Domain: Months 1, 3, 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The general health scale consists of 5 items including a rating of health and 4 items addressing the respondent's view and expectations of his or her health. The domain scores were scored using the US 1998 general population norms. The resulting norm-based T-scores for both the SF36 version 2 & SF36 health domain scales & component summary measures have means of 50 & standard deviations of 10. A higher general health domain score represents better general health perceptions. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
T-scores
  Month 1 (n=128,128,NA,NA,129) | 3.24 (0.529) | 3.74 (0.535) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.29 (0.527)
  Month 3 (n=124,120,NA,NA,117) | 3.67 (0.639) | 3.92 (0.651) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.45 (0.651)
  Month 6 (n=121,111,56,56,NA) | 3.88 (0.695) | 4.46 (0.719) | 6.00 (1.010) | 5.34 (1.010) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

25. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2, Acute Components (SF-36v2 Acute): Vitality Domain: Months 1, 3, 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 4-item measure of vitality captures a broad range of subjective evaluations of well-being from feelings of tiredness and being worn out to feeling full of energy all or most of the time. The domain scores were scored using the US 1998 general population norms. The resulting norm-based T-scores for both the SF36 version 2 & SF36 health domain scales & component summary measures have means of 50 & standard deviations of 10. A higher vitality domain score represents better vitality. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
T-scores
  Month 1 (n=128,128,NA,NA,129) | 4.52 (0.678) | 4.30 (0.684) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 1.73 (0.674)
  Month 3 (n=124,120,NA,NA,117) | 4.95 (0.828) | 4.75 (0.842) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.41 (0.843)
  Month 6 (n=122,111,56,56,NA) | 5.94 (0.859) | 5.15 (0.894) | 5.75 (1.256) | 7.06 (1.256) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

26. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2, Acute Components (SF-36v2 Acute): Social Functioning Domain: Months 1, 3, 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 2-item social functioning scale assesses health-related effects on quantity and quality of social activities. The domain scores were scored using the US 1998 general population norms. The resulting norm-based T-scores for both the SF36 version 2 & SF36 health domain scales & component summary measures have means of 50 & standard deviations of 10. A higher social functioning domain score represents better social functioning. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
T-scores
  Month 1 (n=128,129,NA,NA,129) | 4.93 (0.748) | 4.92 (0.754) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.33 (0.744)
  Month 3 (n=124,120,NA,NA,117) | 6.25 (0.844) | 5.46 (0.861) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.89 (0.861)
  Month 6 (n=122,112,56,56,NA) | 5.92 (0.896) | 5.58 (0.930) | 5.96 (1.309) | 7.90 (1.305) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

27. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2, Acute Components (SF-36v2 Acute): Role-emotional Domain: Months 1, 3, 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 3-item role-emotional scale assesses mental health-related role limitations in terms of a) time spent in work or other usual activities; b) amount of work or activities accomplished; c) care with which work or other activities were performed. All 3 items are answered on a 5-point scale. The domain scores were scored using the US 1998 general population norms. The resulting norm-based T-scores for both the SF36 version 2 & SF36 health domain scales & component summary measures have means of 50 & standard deviations of 10. A higher role-emotional domain score represents better role-emotional functioning. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 125 | 130 | 64 | 65 | 129
T-scores
  Month 1 (n=125,128,NA,NA,129) | 4.44 (0.894) | 3.64 (0.892) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 3.25 (0.878)
  Month 3 (n=121,120,NA,NA,117) | 5.44 (0.998) | 4.84 (1.003) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 3.85 (1.002)
  Month 6 (n=119,111,56,56,NA) | 6.17 (1.010) | 5.69 (1.040) | 7.05 (1.461) | 8.00 (1.455) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

28. Secondary Outcome: Change From Baseline in the Short-Form-36 Health Survey Version 2, Acute Components (SF-36v2 Acute): Mental Health Domain: Months 1, 3, 6
Description: The SF-36v2 acute is a 36-item measure that evaluates 8 domains: physical functioning, role physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. The 5-item mental health scale includes 1 or more items from each of 4 major mental health dimensions: anxiety, depression, loss of behavioral/emotional control, and psychological well-being. All items are answered on a 5-point scale. The domain scores were scored using the US 1998 general population norms. The resulting norm-based T-scores for both the SF36 version 2 & SF36 health domain scales & component summary measures have means of 50 & standard deviations of 10. A higher mental health domain score represents better mental health functioning. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: T-scores
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
T-scores
  Month 1 (n=128,128,NA,NA,129) | 3.80 (0.737) | 4.41 (0.743) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 1.73 (0.732)
  Month 3 (n=124,120,NA,NA,117) | 4.36 (0.852) | 4.11 (0.867) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.11 (0.868)
  Month 6 (n=122,112,56,56,NA) | 4.38 (0.854) | 4.98 (0.884) | 5.06 (1.245) | 5.67 (1.241) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

29. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Mobility: Months 1, 3, 6
Description: The EQ-5D is a descriptive system of health-related quality of life states consisting of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take 1 of 3 responses. The responses record 3 levels of severity (no problems/some or moderate problems/extreme problems) within a particular EQ-5D dimension. Standard vertical 0 to 100 mm VAS (similar to a thermometer) for recording an individual's rating for their current health-related quality of life state, with a higher value representing better health status. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
Units on a scale
  Month 1 (n=128,128,NA,NA,129) | -0.15 (0.035) | -0.10 (0.036) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.08 (0.035)
  Month 3 (n=124,120,NA,NA,117) | -0.17 (0.038) | -0.15 (0.039) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.05 (0.039)
  Month 6 (n=122,112,56,55,NA) | -0.15 (0.040) | -0.15 (0.042) | -0.23 (0.059) | -0.32 (0.059) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

30. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Self-Care: Months 1, 3, 6
Description: as for outcome 29
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 127 | 130 | 64 | 65 | 129
Units on a scale
  Month 1 (n=127,128,NA,NA,129) | -0.11 (0.039) | -0.14 (0.039) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.03 (0.038)
  Month 3 (n=122,120,NA,NA,117) | -0.15 (0.039) | -0.15 (0.040) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.04 (0.039)
  Month 6 (n=120,112,56,55,NA) | -0.19 (0.040) | -0.15 (0.042) | -0.19 (0.058) | -0.17 (0.059) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

31. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Usual Activities: Months 1, 3, 6
Description: as for outcome 29
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
Units on a scale
  Month 1 (n=128,128,NA,NA,129) | -0.22 (0.039) | -0.19 (0.039) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.17 (0.039)
  Month 3 (n=124,120,NA,NA,117) | -0.23 (0.042) | -0.22 (0.042) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.15 (0.043)
  Month 6 (n=122,112,56,55,NA) | -0.30 (0.047) | -0.25 (0.048) | -0.39 (0.068) | -0.34 (0.068) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

32. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Pain/Discomfort: Months 1, 3, 6
Description: as for outcome 29
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
Units on a scale
  Month 1 (n=128,128,NA,NA,129) | -0.26 (0.038) | -0.25 (0.039) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.11 (0.038)
  Month 3 (n=124,120,NA,NA,117) | -0.32 (0.043) | -0.29 (0.044) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.12 (0.044)
  Month 6 (n=121,112,56,55,NA) | -0.34 (0.045) | -0.31 (0.047) | -0.42 (0.066) | -0.34 (0.067) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

33. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on a Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Anxiety/Depression: Months 1, 3, 6
Description: as for outcome 29
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
Units on a scale
  Month 1 (n=128,128,NA,NA,129) | -0.13 (0.043) | -0.21 (0.043) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.10 (0.042)
  Month 3 (n=124,120,NA,NA,117) | -0.19 (0.044) | -0.20 (0.045) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.12 (0.045)
  Month 6 (n=122,112,56,55,NA) | -0.16 (0.046) | -0.20 (0.048) | -0.17 (0.068) | -0.31 (0.068) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

34. Secondary Outcome: Change From Baseline in Score on EuroQol-5 Dimension Health State Profile (EQ-5D) and Change in Patient's Self-rated Health on Vertical Visual Analogue Scale (VAS) Recorded on the EQ-5D Questionnaire (EQ-VAS): Patient's Health State Today: Months 1, 3, 6
Description: as for outcome 29
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: mm
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
mm
  Month 1 (n=127,128,NA,NA,128) | 9.76 (1.565) | 9.58 (1.574) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 3.59 (1.557)
  Month 3 (n=124,119,NA,NA,117) | 8.62 (1.853) | 12.33 (1.896) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.64 (1.896)
  Month 6 (n=122,112,56,55,NA) | 12.14 (1.870) | 12.63 (1.945) | 15.68 (2.736) | 15.32 (2.748) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

35. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scores: Total Score: Months 1, 3, 6
Description: FACIT-F is a 13-item questionnaire, with each item score ranging from 0 to 4. Three endpoints are derived: change in FACIT-F total score, change in FACIT-F experience domain score, and change in FACIT-F impact domain score. FACIT-F total score (range 0-52) is calculated by summing the 13 items. FACIT-F experience domain score (range 0-20) is calculated by summing 5 items : I feel fatigued, I feel weak all over, I feel listless ("washed out"), I feel tired, and I have energy, while FACIT-F impact domain score (range 0-32) is calculated by summing the remaining 8 items. All responses are added with equal weight to obtain the total score. Higher scores represent better fatigue status. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
Units on a scale
  Month 1 (n=128,129,NA,NA,129) | 6.0 (0.66) | 4.4 (0.67) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 2.2 (0.66)
  Month 3 (n=124,120,NA,NA,117) | 7.0 (0.81) | 5.8 (0.82) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 3.0 (0.82)
  Month 6 (n=122,113,56,56,NA) | 7.1 (0.87) | 6.2 (0.90) | 7.6 (1.28) | 8.5 (1.28) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

36. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scores: Experience Domain Score: Months 1, 3, 6
Description: FACIT-F is a 13-item questionnaire, with each item score ranging from 0 to 4. Three endpoints are derived: change in FACIT-F total score, change in FACIT-F experience domain score, and change in FACIT-F impact domain score. FACIT-F total score (range 0-52) is calculated by summing the 13 items. FACIT-F experience domain score (range 0-20) is calculated by summing 5 items : I feel fatigued, I feel weak all over, I feel listless ("washed out"), I feel tired, and I have energy, while FACIT-F impact domain score (range 0-32) is calculated by summing the remaining 8 items. All responses are added with equal weight to obtain the total score. Higher scores represent better (less) fatigue experience. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
Units on a scale
  Month 1 (n=128,129,NA,NA,129) | 2.7 (0.31) | 2.3 (0.31) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 1.0 (0.30)
  Month 3 (n=124,120,NA,NA,117) | 3.1 (0.38) | 2.6 (0.39) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 1.5 (0.39)
  Month 6 (n=122,113,56,56,NA) | 2.9 (0.40) | 2.8 (0.41) | 3.2 (0.58) | 4.1 (0.58) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

37. Secondary Outcome: Change From Baseline in Functional Assessment of Chronic Illness Therapy Fatigue (FACIT-F) Scores: Impact Domain Score: Months 1, 3, 6
Description: FACIT-F is a 13-item questionnaire, with each item score ranging from 0 to 4. Three endpoints are derived: change in FACIT-F total score, change in FACIT-F experience domain score, and change in FACIT-F impact domain score. FACIT-F total score (range 0-52) is calculated by summing the 13 items. FACIT-F experience domain score (range 0-20) is calculated by summing 5 items : I feel fatigued, I feel weak all over, I feel listless ("washed out"), I feel tired, and I have energy, while FACIT-F impact domain score (range 0-32) is calculated by summing the remaining 8 items. All responses are added with equal weight to obtain the total score. Higher scores represent better (less) fatigue impact on daily functioning. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 128 | 130 | 64 | 65 | 129
Units on a scale
  Month 1 (n=128,129,NA,NA,129) | 3.3 (0.40) | 2.1 (0.41) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 1.2 (0.40)
  Month 3 (n=124,120,NA,NA,117) | 3.9 (0.48) | 3.2 (0.49) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | 1.6 (0.49)
  Month 6 (n=122,113,56,56,NA) | 4.2 (0.52) | 3.5 (0.54) | 4.3 (0.76) | 4.5 (0.76) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

38. Secondary Outcome: Change From Baseline in Score Evaluating Spondylitis Using the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI): Months 1, 3, 6
Description: BASDAI is a validated self-assessment tool used to determine disease activity in participants with ankylosing spondylitis. Utilizing a VAS of 0-10 (0=none and 10=very severe) participants answered 6 questions measuring discomfort, pain, and fatigue. The final BASDAI score averaged the individual assessments for a final score ranging 0-10cm, with higher scores representing more severe ankylosing spondylitis disease activity. n=number of participants evaluable at each visit.
Time Frame: Months 1, 3, 6
Population: All participants who were randomized, received at least 1 dose of study drug with presence of spondylitis at screening and baseline BASDAI score >0 cm, and were evaluable.
Measure: Least Squares Mean (Standard Error); unit: cm
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily | Placebo
Number analyzed (Participants) | 26 | 25 | 10 | 12 | 22
cm
  Month 1 (n=26,25,NA,NA,22) | -2.04 (0.400) | -1.26 (0.412) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -0.34 (0.415)
  Month 3 (n=26,22,NA,NA,19) | -2.26 (0.465) | -1.92 (0.490) | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | NA (NA) — Results for this group are reported under the 'Placebo' treatment arm since participants received only placebo up to 3 months. | -1.00 (0.506)
  Month 6 (n=25,22,8,10,NA) | -2.02 (0.463) | -1.56 (0.489) | -2.26 (0.756) | -3.05 (0.701) | NA (NA) — Results for this group are reported under the 'Placebo/Tofacitinib, 5 or 10 mg, twice daily' treatment arms since participants did not receive placebo beyond 3 months.

ADVERSE EVENTS:
Arm/Group | Tofacitinib, 5 mg Twice Daily | Tofacitinib, 10 mg, Twice Daily | Placebo/Tofacitinib, 5 mg, Twice Daily | Placebo/Tofacitinib, 10 mg, Twice Daily
Serious Adverse Events (participants affected / at risk) | 5/131 | 8/132 | 2/66 | 1/65
Other Adverse Events (participants affected / at risk) | 49/131 | 48/132 | 19/66 | 19/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib, 5 mg Twice Daily (N=131) | Tofacitinib, 10 mg, Twice Daily (N=132) | Placebo/Tofacitinib, 5 mg, Twice Daily (N=66) | Placebo/Tofacitinib, 10 mg, Twice Daily (N=65)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0
Parotitis (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tofacitinib, 5 mg Twice Daily (N=131) | Tofacitinib, 10 mg, Twice Daily (N=132) | Placebo/Tofacitinib, 5 mg, Twice Daily (N=66) | Placebo/Tofacitinib, 10 mg, Twice Daily (N=65)
Diarrhoea (Gastrointestinal disorders) | 10 | 8 | 2 | 2
Nausea (Gastrointestinal disorders) | 5 | 7 | 5 | 4
Bronchitis (Infections and infestations) | 3 | 7 | 1 | 2
Nasopharyngitis (Infections and infestations) | 14 | 12 | 4 | 1
Sinusitis (Infections and infestations) | 3 | 5 | 4 | 2
Upper respiratory tract infection (Infections and infestations) | 12 | 7 | 4 | 7
Dizziness (Nervous system disorders) | 7 | 1 | 0 | 1
Headache (Nervous system disorders) | 10 | 12 | 3 | 4
Hypertension (Vascular disorders) | 8 | 5 | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.